CLINICAL TRIAL: NCT02293603
Title: A Randomized, Double-blind, Placebo-controlled, Phase I Study of the Safety of Multi-vessel Intra-coronary Delivery of Allogeneic Human Cardiosphere-Derived Stem Cells in Patients With Dilated Cardiomyopathy (DCM)
Brief Title: Dilated cardiomYopathy iNtervention With Allogeneic MyocardIally-regenerative Cells (DYNAMIC)
Acronym: DYNAMIC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Capricor Inc. (Industry)
Collaborators: Cedars-Sinai Medical Center (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-1002 (DYNAMIC); R44HL095203 (NIH); NCT01815060 (obsolete NCT alias)
Record Dates: First submitted 2014-11-05; First posted 2014-11-18 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Dilated Cardiomyopathy (DCM); Ischemic Cardiomyopathy; Nonischemic Cardiomyopathy; Heart Failure
Keywords: cardiomyopathy; cardiosphere-derived stem cells; intracoronary infusion; adult stem cells; heart disease; ventricular dysfunction; pathological processes; cardiovascular diseases; heart failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Cardiomyopathies; Heart Diseases; Ventricular Dysfunction; Pathologic Processes; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogeneic Cardiosphere-Derived Cells (Experimental): The Phase I study consists of a Phase Ia portion and a Phase Ib portion. The Phase Ia portion (N=14 subjects) consists of an open-label, single-arm, study design. The potentially conducted Phase Ib portion of the study (N=28 subjects) consists of a double-blind, randomized, placebo-controlled study design.
  The Phase Ia portion is an open-label, dose escalation of Allogeneic Cardiosphere-Derived Cells (CDCs).
  Interventions: Biological: Allogeneic Cardiosphere-Derived Cells (CDCs)
- Placebo (Placebo Comparator): The placebo study arm only applies to the Phase Ib portion of the study design. The Phase Ia portion (N=14 subjects) consists of an open-label, single-arm, study design. The potentially conducted Phase Ib portion of the study (N=28 subjects) consists of a double-blind, randomized, placebo-controlled study design.
  Interventions: Biological: Allogeneic Cardiosphere-Derived Cells (CDCs)

INTERVENTIONS:
Biological: Allogeneic Cardiosphere-Derived Cells (CDCs) — Intracoronary delivery of CAP-1002 or placebo
  Other Names: CAP-1002

SUMMARY:
To determine the safety profile of CAP-1002 administered by multi-vessel intracoronary infusion in subjects with DCM. The study will further explore safety and exploratory efficacy endpoints of CAP-1002.

DETAILED DESCRIPTION:
Eligible subjects will undergo sequential intracoronary infusion of CAP-1002 or placebo in up to three coronary arteries supplying three major cardiac territories to the heart (anterior, lateral, inferior/posterior). After completion of the screening procedures, Phase Ia subjects will receive CAP-1002 administered via intracoronary infusion in a dose escalation, stepwise manner. Phase Ia subjects will be followed at Week 2 and at Months 1, 2, 3, 6 and 12 after CAP-1002 infusion. The first fourteen (14) subjects will receive intracoronary infusion of CAP-1002 in an open-label fashion (Phase Ia). Once all 14 subjects in the Phase Ia have reached the primary safety endpoint (1 month visit), the DSMB will conduct a review of the Phase Ia data and recommend whether to proceed with enrollment of the next 28 subjects in the Phase Ib.

ELIGIBILITY:
Major Inclusion Criteria:

1. DCM with left ventricular ejection fraction (LVEF) ≤ 35% as determined by a historical TTE within the previous 6 months
2. New York Heart Association (NYHA) Class III or ambulatory Class IV heart failure
3. Use of evidence based medical-therapy (beta-blockers, ACE-inhibitors/angiotensin receptor blockers, aldosterone antagonist) and with or without device-therapy (Implantable cardioverter-defibrillator or cardiac resynchronizing therapy), in accordance with the ACC/AHA guidelines for the management of heart failure, for at least three months prior to enrollment or documented contraindication or intolerance or patient preference
4. Coronary anatomy suitable for Investigational Product (IP) infusion, as determined by the Eligibility Committee (a team of cardiology experts)
5. Ability to provide informed consent and follow-up with protocol procedures
6. Screening cardiac CT left ventriculogram ejection fraction <40% with left ventricular dilatation
7. Age ≥ 18 years

Major Exclusion Criteria:

1. Diagnosis of active myocarditis
2. Immunologic incompatibility with all available Master Cell Banks (MCBs) by single-antigen bead (SAB) serum antibody profiling
3. Left Ventricular Assist Devices (LVAD) or those actively in the process of acquiring one
4. Recent placement of a cardiac pacemaker and/or resynchronization pacing therapy within the past three months or those actively in the process of acquiring one
5. History of sustained ventricular tachycardia (VT) requiring cardiopulmonary resuscitation (with the exception of subjects who subsequently received an ICD)
6. Non-cardiovascular disease with life expectancy of < 3 years
7. Known hypersensitivity to contrast agents
8. Estimated glomerular filtration rate (GFR) < 50 mL/min
9. Active infection not responsive to treatment
10. Active allergic reactions, connective tissue disease or autoimmune disorders
11. History of cardiac tumor, or cardiac tumor demonstrated on screening
12. History of previous stem cell therapy
13. History of treatment with immunosuppressive agents, including chronic systemic corticosteroids, biologic agents targeting the immune system, anti-tumor and anti-neoplastic drugs or anti-vascular endothelial growth factor (VEGF) within 6 months prior to enrollment (not including drug eluting coronary stents)
14. History of receipt of chemotherapeutic agents known to be implicated in cardiac dysfunction [Adriamycin, trastuzumab (Herceptin)]
15. Known moderate-severe aortic stenosis/insufficiency or severe mitral stenosis/regurgitation
16. Participation in an on-going protocol studying an experimental drug or device
17. Current active alcohol or drug abuse or inability to comply with protocol-related procedures
18. Pregnant/nursing women and women of child-bearing potential without use of active and highly reliable contraception
19. Known history of Human Immunodeficiency Virus (HIV) infection
20. Known history of chronic viral hepatitis
21. Abnormal liver function (serum glutamic pyruvic transaminase (SGPT) > 10 times the upper reference range) and/or abnormal hematology (hematocrit < 25%, white blood cells (WBC) < 3000 µl, platelets < 100,000 µl) studies without a reversible, identifiable cause
22. Evidence of tumor on screening of chest/abdominal/pelvic (body) CT scan
23. Any prior organ transplant
24. Being actively listed for, or under active consideration (i.e., work-up) for, a solid organ transplant of any kind
25. Known hypersensitivity to bovine products
26. Known hypersensitivity to dimethyl sulfoxide (DMSO)
27. Any malignancy within past 2 years (except for in-situ non-melanoma skin cancer and in-situ cervical cancer)
28. Any prior radiation therapy/treatment to the chest
29. Uncontrolled diabetes (HbA1 >9.0)
30. Any condition or other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that experience new TIMI flow 0-2 or TIMI myocardial perfusion grade (TMPG) 0-2. | Intraprocedural
Proportion of subjects that experience acute myocarditis, possibly attributable to CAP-1002. In order to be considered related to CAP-1002, humoral or cellular or immune reaction specific to CAP-1002 must also be documented. | Within one month of intracoronary infusion
Proportion of subjects that experience ventricular tachycardia or ventricular fibrillation resulting in death, appropriate discharge of an ICD or requiring medical intervention. | During or within 72 hours of intracoronary infusion
Proportion of subjects that experience sudden unexpected death occurring within one hour of symptom onset, or un-witnessed death in a person previously observed to be well within the preceding 24 hours without an identified cause. | During or within 72 hours of intracoronary infusion
Proportion of subjects that experience major adverse cardiac events (MACE), including death, non-fatal myocardial infarction and re-hospitalization for cardiovascular event (including heart failure hospitalizations). | During or within 72 hours of intracoronary infusion

SECONDARY OUTCOMES:
Acute myocarditis possibly attributable to CAP-1002. In order to be considered related to CAP-1002, humoral or cellular immune reaction specific to CAP-1002 must also be documented. | During the six & twelve month follow-up period
Ventricular tachycardia or ventricular fibrillation resulting in death or requiring medical intervention or appropriate discharge of an ICD. | During the six & twelve month follow-up period
Sudden unexpected death defined as occurring within one hour of symptom onset, or unwitnessed death in a person previously observed to be well within the preceding 24 hours without an identified cause. | During the six & twelve month follow-up period
Major adverse cardiac events (MACE), including death, non-fatal myocardial infarction, hospitalization for cardiovascular event, emergency room treatment for heart failure, left ventricular assist device or heart transplant. | During the six & twelve month follow-up period
Any hospitalization due to a cardiovascular cause or related to CAP-1002 (or placebo in Phase Ib). | During the six & twelve month follow-up period
Any inter-current cardiovascular illness or one related to CAP-1002 (or placebo in Phase Ib) which prolongs hospitalization. | During the six & twelve month follow-up period
Development of, or an increase in the frequency of, VT with a duration of 30 seconds or longer ascertained by protocol-mandated ECG ambulatory monitoring. | During the six & twelve month follow-up period
Development of increased anti-Human Leukocyte Antigen (HLA) antibody levels with development of sensitization to HLA antigens specific to the CAP-1002 CDC donor at immunologically significant titers. | During the six & twelve month follow-up period
Total number of appropriate ICD firings. | During the six & twelve month follow-up period
Peak elevation in troponin and CKMB levels following CAP-1002 or placebo infusion. | Through Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra (Raj) Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center, Heart Institute; Deborah Ascheim, MD, Study Director — Capricor Inc.
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- See also: Capricor's website — http://capricor.com/